CLINICAL TRIAL: NCT02138591
Title: Therapeutic Benefit of Preoperative Supplemental Vitamin D in Patients Undergoing Major Surgical Procedures.
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: University of Missouri, Kansas City (Other)
Collaborators: Truman Medical Center (Other)
Responsible Party: Principal Investigator, Dustin Neel, Co-Principal Investigator, University of Missouri, Kansas City
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 14-149
Record Dates: First submitted 2014-04-09; First posted 2014-05-14 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Vitamin d Deficiency
Keywords: vitamin d deficiency; cathelicidin antimicrobial peptide; resistin, human; protein, human; 1,25-dihydroxy-16,23-diene vitamin D3; Cholecalciferol; Nutritional Status; length of stay
MeSH Terms: conditions — Vitamin D Deficiency; Muscle Cramp | interventions — Phlebotomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D3 (Experimental): Vitamin D3 (cholecalciferol) 50,000 IU by mouth daily for each of the five days prior to surgery.
  Blood draw pre-operatively Blood draw post-operative Day 1 Blood draw post-operative Day 2
  Interventions: Procedure: Blood draw pre-operatively; Procedure: Blood draw post-operative Day 1; Procedure: Blood draw post-operative Day 2
- Placebo pill (Placebo Comparator): Placebo pill by mouth daily for each of the five days prior to surgery. Blood draw pre-operatively Blood draw post-operative Day 1 Blood draw post-operative Day 2
  Interventions: Procedure: Blood draw pre-operatively; Procedure: Blood draw post-operative Day 1; Procedure: Blood draw post-operative Day 2

INTERVENTIONS:
Procedure: Blood draw pre-operatively — Pre-Operative blood draw of approximately 32ml will check the following: Vitamin D (25-OHD), Calcium, Cathelicidin and Resistin levels in the blood.
  Other Names: Venipuncture
Procedure: Blood draw post-operative Day 1 — Blood draw of approximately 32ml to check the following: Vitamin D (25-OHD), Calcium, Cathelicidin and Resistin levels in the blood.
  Other Names: Venipuncture
Procedure: Blood draw post-operative Day 2 — Blood draw of approximately 32ml to check the following: Vitamin D (25-OHD), Calcium, Cathelicidin and Resistin levels in the blood.
  Other Names: Venipuncture

SUMMARY:
Vitamin D (Vitamin D) deficiency is very common. We recently showed that 97% of 204 patients admitted to Truman Medical Center were Vitamin D deficient (<30 ng/ml). However, the consequences of Vitamin D deficiency, particularly with respect to infection, are not well understood. It is known that production of cathelicidin, an important antimicrobial peptide, is critically dependent upon Vitamin D. It is also established that levels of cathelicidin correlate inversely with urinary tract infection risk. We hypothesize that restoration of Vitamin D levels to normal in patients undergoing major surgery will result in significant decreases in levels of perioperative infections due to restoration of normal levels of circulating Vitamin D, which in turn will elevate cathelicidin levels. As an initial test of this hypothesis, we propose a double-blind, prospective, randomized study of pre-operative Vitamin D supplementation. Fifty subjects undergoing surgery will receive daily Vitamin D3 (50,000 IU) for five days pre-operatively, with controls receiving placebo. Levels of Vitamin D, calcium, cathelicidin, and the pro-inflammatory protein resistin, will be monitored before Vitamin D supplementation (pre-operatively) and after Vitamin D supplementation (post-operative days 1 and 2). The effect of these changes should be to decrease the incidence of infectious complications. We expect to observe Vitamin D levels increase to normal, and cathelicidin levels become elevated. We expect to see increased levels of resistin in patients developing infections. This study will provide strong pilot evidence for future NIH funding.

DETAILED DESCRIPTION:
The long term goal in our research is to develop and implement effective, evidence-and mechanism-based interventions to improve outcomes for surgical and trauma patients. Of potential importance, findings from our own recent pilot studies have established that > 95% of patients seen at Truman Medical Center (TMC) are seriously Vitamin D deficient with plasma levels significantly lower than normal. Our objective in this application, therefore, is to assess the short term therapeutic benefit of high dose Vitamin D in patients admitted to TMC for elective major abdominal surgery. We propose to measure plasma Vitamin D and Calcium levels before supplementation (pre-operatively), and after supplementation (post-operatively), and monitor the biomarker proteins cathelicidin and resistin at the same times. Data on Vitamin D levels will be used to assess direct biochemical effects. Measurement of cathelicidin levels will provide additional information. Since Vitamin D has been shown to induce increased expression of this antimicrobial protein. Monitoring of circulating levels of resistin provides a highly sensitive early measure of infection (unpublished observations). Calcium levels will also be monitored since there is a significant chance that pre-operative calcium levels will be low in some patients, and that supplementation with vitamin D may increase the calcium level.

Measures of secondary clinical outcomes will include length of hospital stay and incidence of post-operation infection. Our central hypothesis is that, relative to patients receiving peri-operative standard of care, patients receiving 250,000 units of Vitamin D pre-operatively will manifest levels of Vitamin D to within the normal range and will have elevated levels of cathelicidin. We further hypothesize that patients receiving Vitamin D will have reduced incidence of infection, which will correlate with lower levels of resistin, and will exhibit trends toward shorter hospital stay. Our proposed specific aims are:

Specific Aim #1: Determine biochemical consequences of Vitamin D supplementation in elective surgery patients We hypothesize that preoperative supplementation with high dose Vitamin D will result in levels of Vitamin D in treated patients within the normal range, corresponding with significant increases in plasma levels of cathelicidin, relative to control patients receiving standard of care.

Specific Aim # 2: Evaluate clinical benefits of Vitamin D supplementation in post-elective surgery patients We postulate that patients given Vitamin D will trend toward lower rates of post-surgery infection, as evidenced by the absence of circulating resistin and decreased detection of pulmonary or wound-site infection, and will have shorter hospital stays relative to patients receiving standard of care.

It is our expectation that, at the completion of this pilot study, we will have provided strong evidence that plasma levels of Vitamin D, as measured by 25-OHD, can be reproducibly raised to normal levels as measured in post-surgery patients and that the administered Vitamin D will have detectable biochemical benefits. We further expect that, while the power of the proposed study will not be sufficient for statistically valid results, there will be trends toward clinical benefits in Vitamin D treated patients. Collectively, these findings would provide strong evidence to support feasibility of an NIH-supported Phase I trial to assess Vitamin D benefits in surgery and/or trauma.

ELIGIBILITY:
Inclusion Criteria:

* English Speaking
* Age 18 years or older
* Patient undergoing major elective surgery with planned open abdominal incisions, and planned hospitalization of two days or longer.

Exclusion Criteria:

* Pregnant
* Non-English Speaking
* Chronic severe kidney disease (Stage III, IV, V)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in Vitamin D level as measured as 25-OHD level | Pre-operatively, Post-operative Day 1 and Postoperative Day 2
  Change in Vitamin D level from Pre-Operatively to Post-Operative Day 1 and Post-Operative Day 2

SECONDARY OUTCOMES:
Change in Resistin level in the blood | Pre-operatively, Post-operative Day 1, Post-operative Day 2
  Change in Resistin level from Pre-Operatively to Post-Operative Day 1 and Post-Operative Day 2
Change in Cathelicidin level in the blood | Pre-operatively, Post-operative Day 1, Post-operative Day 2
  Change in Cathelicidin level from Pre-Operatively to Post-Operative Day 1 and Post-Operative Day 2
Change in Calcium Level in the blood | Pre-operatively, Post-operative Day 1, Post-operative Day 2
  Change in Calcium level from Pre-Operatively to Post-Operative Day 1 and Post-Operative Day 2

CONTACTS AND LOCATIONS:
Overall Officials: Charles Van Way III, M.D., Study Director — Truman Medical Center and University of Missouri Kansas City; Dustin Neel, MD, Principal Investigator — Truman Medical Center and University of Missouri Kansas City
Locations (1):
- Truman Medical Center Hospital Hill, Kansas City, Missouri, United States

REFERENCES:
- [Background] Flynn L, Zimmerman LH, McNorton K, Dolman M, Tyburski J, Baylor A, Wilson R, Dolman H. Effects of vitamin D deficiency in critically ill surgical patients. Am J Surg. 2012 Mar;203(3):379-82; discussion 382. doi: 10.1016/j.amjsurg.2011.09.012. Epub 2011 Dec 28. PMID 22206852
- [Background] Bacon CJ, Gamble GD, Horne AM, Scott MA, Reid IR. High-dose oral vitamin D3 supplementation in the elderly. Osteoporos Int. 2009 Aug;20(8):1407-15. doi: 10.1007/s00198-008-0814-9. Epub 2008 Dec 20. PMID 19101755
- [Background] von Restorff C, Bischoff-Ferrari HA, Theiler R. High-dose oral vitamin D3 supplementation in rheumatology patients with severe vitamin D3 deficiency. Bone. 2009 Oct;45(4):747-9. doi: 10.1016/j.bone.2009.06.012. Epub 2009 Jun 17. PMID 19539796
- [Background] Amrein K, Sourij H, Wagner G, Holl A, Pieber TR, Smolle KH, Stojakovic T, Schnedl C, Dobnig H. Short-term effects of high-dose oral vitamin D3 in critically ill vitamin D deficient patients: a randomized, double-blind, placebo-controlled pilot study. Crit Care. 2011;15(2):R104. doi: 10.1186/cc10120. Epub 2011 Mar 28. PMID 21443793
- [Background] Serrone R, Loveless B, Frankel E, Ross V, Geehan D, Van Way, CW III. vitamin D Deficiency in Patients Admitted to a Midwestern Urban Hospital. Poster presentation at Clinical Nutrition Week, American Society of Parenteral and Enteral Nutrition, Phoenix, AZ, 2013
- [Background] Braun AB, Litonjua AA, Moromizato T, Gibbons FK, Giovannucci E, Christopher KB. Association of low serum 25-hydroxyvitamin D levels and acute kidney injury in the critically ill. Crit Care Med. 2012 Dec;40(12):3170-9. doi: 10.1097/CCM.0b013e318260c928. PMID 22975885
- [Background] Schwalfenberg GK. A review of the critical role of vitamin D in the functioning of the immune system and the clinical implications of vitamin D deficiency. Mol Nutr Food Res. 2011 Jan;55(1):96-108. doi: 10.1002/mnfr.201000174. Epub 2010 Sep 7. PMID 20824663
- [Background] Vieth R. Vitamin D supplementation, 25-hydroxyvitamin D concentrations, and safety. Am J Clin Nutr. 1999 May;69(5):842-56. doi: 10.1093/ajcn/69.5.842. PMID 10232622
- [Background] Ilahi M, Armas LA, Heaney RP. Pharmacokinetics of a single, large dose of cholecalciferol. Am J Clin Nutr. 2008 Mar;87(3):688-91. doi: 10.1093/ajcn/87.3.688. PMID 18326608
- [Background] Gombart AF, Bhan I, Borregaard N, Tamez H, Camargo CA Jr, Koeffler HP, Thadhani R. Low plasma level of cathelicidin antimicrobial peptide (hCAP18) predicts increased infectious disease mortality in patients undergoing hemodialysis. Clin Infect Dis. 2009 Feb 15;48(4):418-24. doi: 10.1086/596314. PMID 19133797
- [Background] White JH. Vitamin D as an inducer of cathelicidin antimicrobial peptide expression: past, present and future. J Steroid Biochem Mol Biol. 2010 Jul;121(1-2):234-8. doi: 10.1016/j.jsbmb.2010.03.034. Epub 2010 Mar 17. PMID 20302931
- [Background] Jeng L, Yamshchikov AV, Judd SE, Blumberg HM, Martin GS, Ziegler TR, Tangpricha V. Alterations in vitamin D status and anti-microbial peptide levels in patients in the intensive care unit with sepsis. J Transl Med. 2009 Apr 23;7:28. doi: 10.1186/1479-5876-7-28. PMID 19389235
- [Background] van der Does AM, Bergman P, Agerberth B, Lindbom L. Induction of the human cathelicidin LL-37 as a novel treatment against bacterial infections. J Leukoc Biol. 2012 Oct;92(4):735-42. doi: 10.1189/jlb.0412178. Epub 2012 Jun 13. PMID 22701042